CLINICAL TRIAL: NCT00956150
Title: Bacterial Overgrowth Associated With Chronic Multisymptom Illness Complex
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry C. Lin, MD (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Henry C. Lin, MD, Henry C. Lin, MD, New Mexico VA Healthcare System
Organization: New Mexico VA Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRRC 07-155
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Gulf War Syndrome
Keywords: Chronic Multisymptom Complex; Small Intestinal Bacterial Overgrowth; Gulf War Syndrome; Chronic Multisymptom Illness Complex
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 60 GWS Rifaximin (Active Comparator)
  Interventions: Procedure: Lactulose Breath Test; Drug: Rifaximin
- 60 GWS Placebo (Placebo Comparator)
  Interventions: Procedure: Lactulose Breath Test; Drug: Placebo
- Healthy Control (Experimental): Patient is a healthy control and will not be on study intervention. Asked to perform Lactulose Breath Test to compare results with GWS patients.
  Interventions: Procedure: Lactulose Breath Test

INTERVENTIONS:
Procedure: Lactulose Breath Test — Test will begin with a baseline breath sample followed by ingestion of 10g of lactulose (Xactdose, South Beloit, IL) in 100ml of water. Breath samples will be collected every 15 min for 180 min. Gas samples will be analyzed for hydrogen and methane using a gas chromatograph (Model SC, Quintron Instruments, Milwaukee, WI).
Drug: Rifaximin — Rifaximin 600 mg three times a day by mouth (TID PO) x 10 days
  Arms: 60 GWS Rifaximin
Drug: Placebo — Placebo TID PO x 10 days
  Arms: 60 GWS Placebo

SUMMARY:
The adverse impact of Gulf War Syndrome (GWS) on the health of veterans and on the resources of the VA Healthcare System underscores the need to resolve its underlying cause. In response, the investigators propose to investigate the central hypothesis that gut bacteria may be responsible for symptoms associated with GWS. The investigators will enroll a total of 120 patients with GWS and 90 healthy controls.

DETAILED DESCRIPTION:
The investigator will assess the prevalence and role of abnormal gut microbial fermentation among Veterans with GWS and investigate the efficacy of diagnostic and treatment strategies directed at indigenous gut microbes in the management of GWS.

ELIGIBILITY:
Inclusion Criteria:

* Gulf War Veterans meeting the 1994 Centers for Disease Control and Prevention (CDC) criteria for the diagnosis of Chronic Fatigue Syndrome(CFS), i.e > six months of one or more symptoms from at least two of the following three clusters: general fatigue, mood and cognitive abnormalities, and musculoskeletal pain
* Must be under the care of a primary physician and have had a previous diagnosis of Gulf War-related illness or GWS and have medical records documenting investigations to rule out other causes of fatigue
* Minimum of the following laboratory screening tests: complete blood count with leukocyte differential, erythrocyte sedimentation rate, serum electrolytes, calcium, glucose, blood urea nitrogen, creatinine,urinalysis, and thyroid function tests
* Subjects must also have a GI consult first as part of routine care to confirm eligibility and availability
* Patients with Irritable Bowel Syndrome (IBS), fibromyalgia (FM), anxiety or depression will not be excluded, but will be identified for subgroup analysis
* Healthy controls will be screened with complete blood count (CBC) and comprehensive metabolic panel to confirm eligibility

Exclusion Criteria:

* History of peptic ulcer, inflammatory bowel disease, diabetes, cirrhosis, rheumatoid arthritis, lupus, narcotic dependence,celiac disease, tropical sprue, bowel resection(including gastric, small bowel or colon; but gallbladder surgery or appendectomy are NOT exclusion criteria)
* Patients with chronic illness (HIV, tuberculosis)
* Pregnant or breast-feeding, psychotic depression, bipolar disorder, schizophrenia, eating disorders
* Healthy subjects will be excluded if their questionnaire indicated abnormal symptom profile

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2009-04; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
To compare the pattern of bacterial gas excretion in breath among Veterans with Gulf War Syndrome vs. Controls using Lactulose Breath Test | every 15 minutes for 180 minutes
To determine the response to antibiotic treatment in Gulf War Syndrome patients. | Two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- New Mexico VA Healthcare System, Albuquerque, New Mexico, United States